CLINICAL TRIAL: NCT04208646
Title: A Multicenter, Randomized, Double-blind, Controlled Phase II Trial of Allogenic Adipose Tissue-Derived Mesenchymal Progenitor Cells (AlloJoin®) for the Treatment of Knee Osteoarthritis
Brief Title: Allogenic Adipose Tissue-Derived Mesenchymal Progenitor Cells for the Treatment of Knee Osteoarthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai AbelZeta Ltd. (Industry)
Collaborators: RenJi Hospital (Other); Shanghai 6th People's Hospital (Other); Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); China-Japan Friendship Hospital (Other); Huashan Hospital (Other); Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CBM-ALAM.1-01
Record Dates: First submitted 2019-12-17; First posted 2019-12-23 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-05

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mesenchymal progenitor cells Dosage 1 (Experimental): Mesenchymal progenitor cells low-dose group
  Interventions: Biological: Mesenchymal progenitor cells
- Mesenchymal progenitor cells Dosage 2 (Experimental): Mesenchymal progenitor cells high-dose group
  Interventions: Biological: Mesenchymal progenitor cells
- No mesenchymal progenitor cells (Placebo Comparator): No mesenchymal progenitor cells
  Interventions: Biological: No mesenchymal progenitor cells

INTERVENTIONS:
Biological: Mesenchymal progenitor cells — Allogenic Adipose tissue-derived mesenchymal progentior cells administrated for intra- articular use
  Arms: Mesenchymal progenitor cells Dosage 1; Mesenchymal progenitor cells Dosage 2
Biological: No mesenchymal progenitor cells — No mesenchymal progenitor cells for intra- articular use
  Arms: No mesenchymal progenitor cells

SUMMARY:
Evaluate the efficacy and safety of Allogenic Adipose Tissue-Derived Mesenchymal Progenitor Cells Therapy

DETAILED DESCRIPTION:
A Multicenter, Randomized, Double-blind, Controlled Phase II Trial of Allogenic Adipose Tissue-Derived Mesenchymal Progenitor Cells (AlloJoin®) Therapy for Knee Osteoarthritis.

This is a multicenter, randomized, double-blinded, phase II clinical trial. Subjects who are with a clinical diagnosis of knee osteoarthritis cartilage defects and will be randomly distributed 1:1:1 to different group after signing the ICF and screening tests. Each group was treated for two cycles. The patients were followed up to 48 weeks after the first treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who understand and voluntarily sign the consent form before this study；
2. According to the diagnostic criteria (American Rheumatology Association, clinical + radiology criteria), patients with knee osteoarthritis are definitely diagnosed；
3. Age: 40-75, males and females；
4. The course of knee osteoarthritis was more than 6 months and less than 10 years;
5. The subjects' WOMAC score was 24-72, and the WOMAC pain score was 7-17 (the WOMAC score at least 48 hours after discontinuation of all painkillers);
6. The Kellgren Lawrence grade (X-ray axial position of knee joint) of subjects was grade II / III;
7. Subjects are generally in good condition and can walk autonomously, except for those who use wheelchairs, walking aids or crutches.

Exclusion Criteria:

1. The subject may be allergic to the main cell preparation components (B vitamins, amino acids and so on).
2. The subject received systemic and / or local treatment with autologous and / or allogeneic mesenchymal progenitor cells.
3. The subject has a BMI of over 30.
4. Laboratory test (any item meets): neutrophil absolute number < 1.0 × 10^9 / L, platelet count < 50 × 10^9 / L, serum albumin < 30g / L, serum creatinine > upper limit of normal value range, total bilirubin、alanine aminotransferase、aspartate aminotransferase > upper limit of 2 times of normal value range.
5. The subject has diseases or symptoms may affect VAS, WOMAC and so on.
6. The subject has serious and poorly controlled concomitant diseases, such as (but not limited to) nervous system, cardiovascular, liver, kidney, gastrointestinal and endocrine diseases, which may prevent the subjects from participating in the study according to the judgment of the researchers.
7. The subject has an history malignant tumour.
8. The subject has connective tissue disease or rheumatoid arthritis、chondropathy、Chondrocalcinosis articularis、 Hemochromatosis、inflammatory arthropathy、avascular necrosis of femoral head、Paget's disease、hemophilic arthropathy、infectional arthritis、Charcot' s disease、villonodular synovitis or synovial chondromatosis.
9. The subject has severe generalized infectious diseases or local knee infection (including skin and intra-articular infection) in the 3 months prior to this trial.
10. According to the researchers,the subject has disease of lower limbs which may be interfered knee evaluation, for example fibromyalgia, osphyalgia, lumbar disc protrusion and so on.
11. The subject had any other coagulation dysfunction caused by acute or chronic diseases, according to the judgment of the researchers, this coagulation dysfunction may endanger the safety of patients and / or affect the judgment of knee joint evaluation indicators.
12. The subject has received arthroscopic surgery or other open surgery related to knee joint operation in the 6 months prior to this trial.
13. The subject has received other intra-articular injections, including but not limited to hyaluronic acid, hormone, PRP, BMP (bone morphogenetic protein) , hypertonic glucose and so on for KOA in the 3 months preceding the trial.
14. The subject has received aminoglucose or chondroitin sulfate within 1 month before the treatment.
15. The subject has used dexamethasone, prednisone, hydrocortisone and other hormones orally / intravenously within 1 month before the treatment.
16. The subject has undergone knee prosthesis or a plan of knee prosthesis within the trial.
17. The subject has contraindication of MRI, included but not only: the subject installed heart pacemaker, defibrillator, heart bracket, heart valve prosthesis, metal clip after aneurysm surgery, drug infusion device implanted in vivo, any electronic device implanted in the body (nerve stimulator, bone growth stimulator) endovascular coil, strainer, ECG monitor, metal suture, shrapnel or sand of body, plate fixation and steel nail after fracture surgery, artificial cochlea, middle ear shift plant, metallic intraocular foreign body etc; the subject is a claustrophobia, critical ill patient and so on.
18. The subject tests positive for: HIV, HBV, HCV and treponema pallidum.
19. The subject has history of alcoholism, drug abuse, or mental illness in the 3 years prior to this trial.
20. The subject has participated in any other clinical trial in the 3 months prior to this trial.
21. The subject (including male subjects) has fertility, sperm donation or egg donation plans during the trial period; the female subject is pregnant, lactating or having a positive pregnancy test.
22. The subject is legally disabled by reference to the law of the people's Republic of China on the protection of disabled persons (April 2008).
23. The subject has any other unsuitable condition (such as factors reducing the follow-up compliance) to be determined by the investigator.

24.The Kellgren Lawrence grade (X-ray axial position of knee joint) of any knee joint of the subjects was grade IV.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2020-05-16 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
WOMAC Score | 24 weeks
  The Western Ontario and McMaster Universities Osteoarthritis Index;0-96 points；96 points mean a worse outcome,will be tested at 24 weeks after the first injection

SECONDARY OUTCOMES:
MRI quantitative analysis of articular cartilage | 24 weeks,48 weeks
  Magnetic Resonance Imaging analysis of articular cartilage, will be tested at 24、48 weeks after the first injection
WOMAC Score | 4、8、12、36、48 weeks
  The Western Ontario and McMaster Universities Osteoarthritis Index;0-96 points；96 points mean a worse outcome, will be tested at 4、8、12、36、48 weeks after the first injection
VAS Score | 4、8、12、24、36、48 weeks
  Visual Analogue Scale/Score；0-10 points；10 points mean a worse outcome,will be tested at 4、8、12、24、36、48 weeks after the first injection
SF-36 | 4、8、12、24、36、48 weeks
  The Medical Outcomes Study 36-Item Short-Form Health Survey;0-100 points；100 points mean a better outcome, will be tested at 4、8、12、24、36、48 weeks after the first injection
Adverse Events and Serious Adverse Events | 0d、1、3、4、8、12、24、25、27、28、36、48 weeks
  AE and SAE, will be assessed at 0d、1、3、4、8、12、24、25、27、28、36、48 weeks
Changes of laboratory test indexes and vital signs | 0d、1、3、4、8、12、24、25、27、28、36、48 weeks
  Vital signs, physical examination, clinical laboratory tests:infectious disease check, blood coagulation test , blood check, urine check, blood biochemical test, immunological examination, tumor screening ,will be tested at 0d、1、3、4、8、12、24、25、27、28、36、48 weeks

OTHER OUTCOMES:
Metabolic index detection | 0、4、8、12、24、36、48 weeks
  Levels of cartilage metabolism and inflammatory biomarkers in serum and urine will be tested at 0、4、8、12、24、36、48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Chunde Bao, Principal Investigator — RenJi Hospital; Changqing Zhang, Principal Investigator — Shanghai 6th People's Hospital; Guochun Wang, Principal Investigator — China-Japan Friendship Hospital; Chengqing Yi, Principal Investigator — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine; Shigui Yan, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University; Weiguo Wan, Principal Investigator — Huashan Hospital; Jinwu Wang, Principal Investigator — Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Locations (7):
- China (7):
  - China-Japan Friendship Hospital, Beijing
  - The Second Affiliated hospital of Zhejiang University School of Medicine, Hangzhou
  - Huashan Hospital Affiliated to Fudan University, Shanghai
  - Shanghai General Hospital, Shanghai
  - Shanghai Jiaotong University School of Medicine, Renji Hospital, Shanghai
  - Shanghai Sixth People's Hospital, Shanghai
  - Shanghai Ninth People's Hospital, Shanghai JiaoTong University School of Medicine, Shanghai